CLINICAL TRIAL: NCT01446042
Title: A 90-Day, Randomized, Dose-Ranging Study, Including Potential Dose Titration, Evaluating the Efficacy and Safety of Intranasal TBS-1 in the Treatment of Male Hypogonadism With Sequential Safety Extension Periods of 90 and 180 Days
Brief Title: Safety and Efficacy of Intranasal TBS-1 Treatment of Male Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBS-1-2011-03
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-03

CONDITIONS: Male Hypogonadism
MeSH Terms: conditions — Eunuchism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TBS-1 - b.i.d. (Experimental): 5.5 mg per nostril of 4.5% TBS-1 BID
  Interventions: Drug: Testosterone
- TBS-1 - t.i.d. (Experimental): 5.5 mg per nostril of 4.5% TBS-1 TID
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Intranasal testosterone
  Arms: TBS-1 - b.i.d.
Drug: Testosterone — Intranasal testosterone
  Arms: TBS-1 - t.i.d.

SUMMARY:
The purpose of this study is to determine the efficacy (based on the pharmacokinetic profile of testosterone) and safety of TBS-1 in the treatment of hypogonadal men

DETAILED DESCRIPTION:
This study is a 4 Period study consists of 16 visits with overnight clinic stays that span over year to help determine the efficacy of TBS-1 gel administered twice daily (b.i.d) and three times daily (t.i.d)

In addition, this study will investigate the safety and tolerability of TBS-1 after 90, 180 and 360 days of treatment.

ELIGIBILITY:
Inclusion Criteria

* Male between 18 and 80 years of age
* Able to understand and provide signed informed consent
* Have 2 fasting morning (0900 h ± 30 min) serum total testosterone levels <300 ng/dL
* Body mass index between 18.5 kg/m2 and 35 kg/m2
* Hemoglobin level > or = 13.0 g/dL
* Screening laboratory assessments within ±15% of the normal range, with the exception of liver function tests (which need to be within the normal range) and HbA1c (which must be <7.0% [9.5 mmol/L]); lipid profile and endocrine profile assessments are also exempt from this range unless the assessments indicate a significant intercurrent illness other than testosterone deficiency
* Ear, nose and throat examination including nasal endoscopy without clinically significant abnormal findings
* Normal prostate for age based on digital rectal exam and a serum PSA <4.0 ng/mL.

Exclusion Criteria

* Significant intercurrent disease of any type, in particular liver, kidney, heart disease, or psychiatric illness
* Hyperparathyroidism, uncontrolled diabetes mellitus, hypothyroidism, or hyperthyroidism (thyroid stimulating hormone should be <1.5 times the upper limit of normal)
* Hematocrit >54% at screening
* History of pituitary or hypothalamic tumors or history of malignancy within the past 5 years, excluding basal cell or squamous cell carcinoma of the skin curatively treated by surgery
* History of nasal surgery, specifically turbinoplasty, septoplasty, rhinoplasty, "nose job," or sinus surgery
* History of nasal fractures within the past 6 months and/or prior nasal fractures that caused a severely deviated anterior nasal septum
* Active allergies, such as rhinitis, rhinorrhea, and nasal congestion
* Mucosal inflammatory disorders, specifically pemphigus or Sjogren's syndrome
* Sinus disease, specifically acute sinusitis, chronic sinusitis, or allergic fungal sinusitis
* History of nasal disorders (eg, polyposis, recurrent epistaxis [>1 nose bleed per month], abuse of nasal decongestants) or sleep apnea
* Use of any form of intranasal medication delivery, specifically nasal corticosteroids and oxymetazoline-containing nasal sprays (eg, Dristan® 12-Hour Nasal Spray)
* History of severe adverse drug reaction or leukopenia
* A known hypersensitivity to lidocaine or any materials that may be used during the study
* History of abnormal bleeding tendencies or thrombophlebitis unrelated to venipuncture or intravenous cannulation
* History of hepatitis B, a positive test for hepatitis B surface antigen, a history of hepatitis C, or a positive test for hepatitis C antibody
* Presence of human immunodeficiency virus infection or antibodies
* History of asthma and ongoing asthma treatment
* History of sleeping problems or a shift worker
* Smoker of >10 cigarettes (or equivalent) per day
* Regular consumption of more than 4 units of alcohol daily (1 unit is defined as 300 mL of beer, 1 glass of wine, or 1 measure of spirit) or difficulty abstaining from alcohol during the 48 hours prior to the 24 hour blood sampling visits
* History or current evidence of abuse of alcohol or any drug substance, licit or illicit, or positive urine drug and alcohol screen
* Treatment with androgen therapy within at least 2 weeks prior to baseline evaluations (subjects on androgen therapy will require a washout period of 4 weeks for depot products administered intramuscularly [eg, testosterone enanthate 200 mg/mL] and 2 weeks for products administered orally or topically [oral, patch, gel, or buccal])
* Current treatment with other androgens (eg, dehydroepiandrosterone [DHEA]), anabolic steroids, or other sex hormones
* Treatment with estrogens, gonadotropin-releasing hormone (GnRH) agonists, or growth hormone within previous 12 months
* Treatment with drugs that interfere with the metabolism of testosterone, such as anastrozole, clomiphene, dutasteride, finasteride, flutamide, ketoconazole, spironolactone, or testolactone
* Treatment with any antihypertensive, antidepressant, tranquilizer, or histamine 2 (H2) receptor blocker that is not part of a stable regimen (stable dose for at least 3 months prior to baseline);
* Poor compliance history or low likelihood of maintaining attendance
* Participation in any other research study during the conduct of this study or 30 days prior to the initiation of this study or blood donation at any time during this study and within the 12 week period prior to screening

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Tkachenko, MD, Study Director — Trimel Pharmaceuticals Corporation
Locations (30):
- United States (30):
  - Alabama Clinical Therapeutics LLC, Birmingham, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Quality of Life Medical Research Center, Tucson, Arizona
  - SC Clinical Research Inc, Garden Grove, California
  - Diablo Clinical Reseach Inc., Walnut Creek, California
  - Innovative Research of West Florida, Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Compass Research East LLC, Oviedo, Florida
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Commonwealth Biomedical Research LLC, Madisonville, Kentucky
  - Regional Urology LLC, Shreveport, Louisiana
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Rochester Clinical Research, Rochester, New York
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center Inc, Mt. Pleasant, South Carolina
  - Austin Center for Clinical Research, Austin, Texas
  - Reseach Across America, Dallas, Texas
  - Centex Research, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Cetero Research, San Antonio, Texas
  - Granger Medical Clinic, West Valley City, Utah
  - National Clinical Research - Norfolk, Norfolk, Virginia
  - National Clinical Research, Richmond, Virginia
  - Capital Clinical Reseach Center, Olympia, Washington
  - Rainier Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Rogol AD, Tkachenko N, Bryson N. Natesto , a novel testosterone nasal gel, normalizes androgen levels in hypogonadal men. Andrology. 2016 Jan;4(1):46-54. doi: 10.1111/andr.12137. Epub 2015 Dec 22. PMID 26695758

RESULTS

PARTICIPANT FLOW:
Groups:
- TBS-1 - b.i.d.: Intranasal testosterone given b.i.d.
- TBS-1 b.i.d./t.i.d: Subjects on b.i.d. who were uptitrated to t.i.d. on Day 45
- TBS-1 - t.i.d.: Intranasal testosterone given t.i.d.
Period: Overall Study
Arm/Group | TBS-1 - b.i.d. | TBS-1 b.i.d./t.i.d | TBS-1 - t.i.d.
Started | 142 | 86 | 78
Completed | 122 | 83 | 69
Not Completed | 20 | 3 | 9
Not completed — Withdrawal by Subject | 12 | 2 | 4
Not completed — Adverse Event | 1 | 0 | 4
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Other reasons | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- TBS-1 - b.i.d./t.i.d.: Subjects on b.i.d. who were uptitrated to t.i.d. on Day 45
- Total: Total of all reporting groups
Arm/Group | TBS-1 - b.i.d. | TBS-1 - b.i.d./t.i.d. | TBS-1 - t.i.d. | Total
Number analyzed (Participants) | 142 | 86 | 78 | 306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 121 | 64 | 61 | 246
  >=65 years | 21 | 22 | 17 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 142 | 86 | 78 | 306
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 142 | 86 | 78 | 306

OUTCOME MEASURES:

1. Primary Outcome: Serum Testosterone Cavg
Description: The percentage of patients with an average serum total testosterone concentration (Cavg) within the normal range (300 to 1050 ng/dL)
Time Frame: 90 days
Population: Per-Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | TBS-1 - b.i.d. | TBS-1 - b.i.d./t.i.d. | TBS-1 - t.i.d.
Number analyzed (Participants) | 102 | 68 | 67
Participants | 76 | 43 | 61

2. Secondary Outcome: Patients With a Certain Serum Total Testosterone Maximum Concentration on Day 90
Description: To determine the efficacy of 4.5% TBS-1 gel, administered 2 or 3 times daily at a dose of 5.5 mg per nostril, in achieving the following serum total testosterone maximum concentration (Cmax) on Day 90:
  * A Cmax (maximum testosterone concentration) value of 1500 ng/dL or more in at least 85% of the participants analyzed
  * A Cmax (maximum testosterone concentration) value of 1800 to 2500 ng/dL in fewer than 5% of participants analyzed
  * No analyzed participants with a Cmax (maximum testosterone concentration) >2500 ng/dL
Time Frame: 90 days
Population: ITT subjects who have a Cmax value at the specified visit.
Measure: Count of Participants; unit: Participants
Arm/Group | TBS-1 - b.i.d. | TBS-1 - b.i.d./t.i.d. | TBS-1 - t.i.d.
Number analyzed (Participants) | 114 | 79 | 59
Participants
  Cmax <=1500 ng/dL | 107 | 77 | 58
  1800 ng/dL <= Cmax <=2500 ng/dL | 6 | 2 | 1
  Cmax >2500 ng/dL | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TBS-1 - b.i.d. | TBS-1 - b.i.d./t.i.d. | TBS-1 - t.i.d.
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/86 | 1/78
Serious Adverse Events (participants affected / at risk) | 2/142 | 1/86 | 2/78
Other Adverse Events (participants affected / at risk) | 65/142 | 40/86 | 46/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBS-1 - b.i.d. (N=142) | TBS-1 - b.i.d./t.i.d. (N=86) | TBS-1 - t.i.d. (N=78)
Internal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament Rapture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TBS-1 - b.i.d. (N=142) | TBS-1 - b.i.d./t.i.d. (N=86) | TBS-1 - t.i.d. (N=78)
Retching (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Chills (General disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 4 | 3
Bronchitis (Infections and infestations) | 2 | 0 | 3
Tooth abscess (Infections and infestations) | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 3
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 2
PSA increased (Investigations) | 0 | 2 | 4
Blood CPK increased (Investigations) | 1 | 2 | 2
Blood pressure increased (Investigations) | 0 | 1 | 2
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 2
Weight increased (Investigations) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Parosmia (Nervous system disorders) | 7 | 3 | 2
Headache (Nervous system disorders) | 2 | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Scab (Skin and subcutaneous tissue disorders) | 3 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes